CLINICAL TRIAL: NCT00632437
Title: Intraoperative Optical Imaging of Brain Function
Status: Withdrawn | Type: Observational
Why Stopped: Terminated due to poor enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0102
Record Dates: First submitted 2008-02-13; First posted 2008-03-10 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Brain Tumor
Keywords: Brain Tumor; Craniotomy Surgery; Brain Function; Intraoperative Optical Imaging; Speckle-Contrast Imaging; Cortical Mapping; Somatosensory Cortex; Cerebral blood flow; CBF; Laser Speckle Contrast Imaging; Multi-Spectral Imaging
MeSH Terms: conditions — Brain Neoplasms | interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Speckle-Contrast Imaging
  Interventions: Procedure: Speckle-Contrast Imaging

INTERVENTIONS:
Procedure: Speckle-Contrast Imaging — Imaging camera scan that uses reflected red light to take pictures of the amount of blood flowing in brain and the amount of oxygen in blood.

SUMMARY:
The goal of this proposal is to test the performance of a novel optical imaging system for real-time quantitative imaging of brain function through multiple hemodynamic measures during neurosurgery.

This pilot study encompasses two sub-aims:

* Evaluate the ability of laser speckle contrast imaging to image cerebral blood flow (CBF) intraoperatively. We will image the changes in CBF in response to somatosensory stimulation. (5 patients).
* Simultaneously image hemoglobin oxygenation, blood volume, blood flow, and cerebral metabolic rate of oxygen (CMRO2) changes during somatosensory stimulation using a combined laser speckle and multi-wavelength reflectance imaging system. (5 patients).

DETAILED DESCRIPTION:
A speckle-contrast imaging camera uses a low-power laser to check brain activity. The imaging camera uses reflected red light to take a special kind of picture of the amount of blood flowing in your brain, and the amount of oxygen in your blood. This is the first time this device has been used in brain surgery.

While "asleep" under anesthesia during an already scheduled surgery, the neurosurgeon will position the microscope to take pictures of the surgery area. The pictures will be taken after the brain is exposed, but before the rest of the surgery takes place. Researchers will shine the red light onto the brain during your surgery. The light will then be seen by the camera.

"Cortical mapping" will done, which is an established procedure used to detect important areas of the brain. Usually, a nerve in the wrist is stimulated with a very small shock of electricity and a response is detected in the brain by an electrode placed on the surface. The electrical shock administered is not dangerous or painful. It will be given while "asleep." For the experimental procedure used in this study, the same stimulation will be used, but the impulse detection will be performed using the speckle-contrast imaging camera. Researchers hope to see if the change in blood flow gives the same information as if the electrode was placed on the brain and used to detect the electricity. Doing both procedures is expected to take no more than 20 minutes. During this time, continual monitoring done by the surgeon and operating room staff.

Your participation in this study will end when the surgery is finished.

The results of this study will not be used by the surgeon during your surgery or any future treatments. These measurements are being done for research only and will not be used by the surgeon to make any decisions about your surgery.

This is an investigational study. This device is investigational and has not been approved by the Food and Drug Administration (FDA), but it has been declared safe by the National Institutes of Health. Up to 10 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Location of planned resection near somatosensory cortex.
2. Planned intraoperative electrocortical mapping.
3. Able to render written informed consent.

Exclusion Criteria:

1. Patients with a hemiparesis graded 3/5 (active movement against gravity) or worse. Unpublished data from MDACC Department of Neurosurgery suggests that cortical mapping is ineffective in these patients because an adequate cortical response is not detected
2. Patients with a vascular malformation within the proximity of the cortex area imaged.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having a brain tumor which is scheduled to be surgically removed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Test performance of novel optical imaging system for real-time quantitative imaging of brain function through multiple hemodynamic measures during neurosurgery | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weinberg, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org